CLINICAL TRIAL: NCT00003324
Title: Prognostic Factors Associated With Successful Omission of Whole Brain Radiotherapy in Patients With 4 or Less Cerebral Metastases Treated With Focal Radiation or Surgery
Brief Title: Radiation Therapy With or Without Surgery in Treating Patients Who Have Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066275; UCLA-HSPC-9710074; UCLA-HSPC-971007401; NCI-G98-1417
Record Dates: First submitted 1999-11-01; First posted 2003-04-25 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Metastatic Cancer
Keywords: tumors metastatic to brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells in a single high dose. Combining radiation therapy with surgery may be a more effective treatment for brain metastases.

PURPOSE: Clinical trial to study the effectiveness of radiation therapy with or without surgery in treating patients who have brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop prognostic factors for patients with brain metastases treated by focal treatment without concurrent whole brain irradiation.
* Determine whether focal treatment without whole brain radiotherapy produces good long-term outcome in patients with four or less cerebral metastases.
* Assess survival, physical and cognitive functioning, and quality of life of patients treated on this protocol.

OUTLINE: Quality of life is assessed using the FACT-BR scale, physical function is assessed using the FIM scale, and cognition is assessed using two brief pencil and paper tests.

Patients receive focal therapy for cerebral metastases by any combination of (1) surgery plus fractionated stereotactic radiotherapy to surgical bed, or (2) single fraction stereotactic radiotherapy by linear accelerator with or without a radiation sensitizer.

Patients are followed at 2 and 10 weeks, then every 3 months for 18 months, then every 6 months for 3 years, then annually. Quality of life is assessed at each followup visit.

Patients suffering intracerebral relapse are offered further focal therapy if they have no more than 3 metastases, no more than 6 lesions over consecutive scans, and continue to have life expectancy of at least 3 months and Karnofsky performance status of 60-100%. Otherwise, relapsed patients are offered whole brain radiotherapy or supportive treatment with steroids, and may also receive stereotactic boost to the new lesions. Patients who have received prior whole brain irradiation will be offered entry into other protocols if eligible or supportive treatment with steroids. Patients are followed as above.

PROJECTED ACCRUAL: At least 60 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy, CT scan, or MRI proven cerebral metastases with known current or previous systemic malignancy OR
* Biopsy proven cerebral metastases other than from small cell lung cancer or lymphoma
* Refused whole brain radiation therapy OR
* Received prior whole brain radiation therapy and ineligible for other relapse protocols
* 18 and over
* Karnofsky 60-100%
* Life expectancy:At least 3 months
* Concurrent steroids allowed

Exclusion Criteria:

* more than four cerebral metastases on MRI scan and suitable for focal treatment with surgery and/or stereotactic radiotherapy with a linear accelerator
* more than 2 weeks since prior focal radiation
* more than 2 weeks since prior focal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 1997-12; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Ford, MD, PhD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Chitapanarux I, Goss B, Vongtama R, Frighetto L, De Salles A, Selch M, Duick M, Solberg T, Wallace R, Cabatan-Awang C, Ford J. Prospective study of stereotactic radiosurgery without whole brain radiotherapy in patients with four or less brain metastases: incidence of intracranial progression and salvage radiotherapy. J Neurooncol. 2003 Jan;61(2):143-9. doi: 10.1023/a:1022173922312. PMID 12622453